CLINICAL TRIAL: NCT05593315
Title: Efficacy of the Combination of General Relaxation (Mindfulness) and Respiratory (Buteyko) Techniques for the Improvement of Poorly Controlled Asthma. The MBA Study
Brief Title: Efficacy of the Combination of Mindfulness and Buteyko Techniques for the Improvement of Poorly Controlled Asthma.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IIBSP-MBA-2022-95
Record Dates: First submitted 2022-10-10; First posted 2022-10-25 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Asthma; Anxiety; Stress
Keywords: Asthma; Anxiety; Stress; Mindfulness; Buteyko
MeSH Terms: conditions — Asthma; Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: A Mindfulness relaxation program and a Buteyko technique respiratory rehabilitation program will be administered individually and weekly, in 10 sessions (5 face-to-face and 5 telematic sessions afterwards).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness and Buteyko techniques (Other): A Mindfulness relaxation program and a Buteyko technique respiratory rehabilitation program will be administered individually and weekly, in 10 sessions (5 face-to-face and 5 telematic sessions afterwards).
  Interventions: Other: Mindfulness and Buteyko techniques

INTERVENTIONS:
Other: Mindfulness and Buteyko techniques — Joint implementation of a general relaxation program and a respiratory rehabilitation program in patients with poorly controlled asthma.

SUMMARY:
Administration of a combined program for general (Mindfulness) and respiratory (Buteyko technique) relationship in patients with poorly controlled asthma and anxiety/stress to determine if it provides an improvement in current control and future risk of asthma.

DETAILED DESCRIPTION:
A Mindfulness relaxation program and a Buteyko technique respiratory rehabilitation program will be administered individually and weekly, in 10 sessions (5 face-to-face and 5 telematic sessions afterwards). Patients will be visited 4 times (at inclusion, one month, 6 months and 12 months after the double intervention), where data on asthmatic morbidity, pulmonary function (spirometry), bronchial inflammation (FENO) will be collected and some questionnaires will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of poorly controlled asthma
* In treatment with a combination of ICS/LABA at medium doses
* Anxiety and/or functional dyspnea
* Attended in the outpatient consultations of the Asthma Unit of the Pneumology and Allergy Service of the Hospital de la Santa Creu i Sant Pau in Barcelona

Exclusion Criteria:

* Severe asthma exacerbation in the last 30 days
* Severe disabling comorbidity
* Severe psychiatric illness
* Inability to complete questionnaires.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
% patients with changed asthma control | 1 year
  Changes in asthma symptoms measured with the asthma control test (minimum 5 as worse value; maximum 25, as the best value)
Changes in asthma exacerbation | 1 year
  Changes in asthma exacerbation measured by number of hospital admissions and medical treatments received

SECONDARY OUTCOMES:
Anxiety | 1 year
  Improvement of the anxiety level measured with the test hospital anxiety and depression scale (minimum 0 as the best value, maximum 42 as the worst value)
Functional dyspnea | 1 year
  Changes in functional dyspnea measured with the test Nijmegen (minimum 0 as the worst value, maximum 64 as the worst value)
Pulmonary function | 1 year
  Changes in pulmonary function with spirometry (Forced Expiratory Volume in 1 Second and forced vital capacity)
Bronchial inflammation | 1 year
  Changes in bronchial inflammation with FENO
Therapeutic adherence of patients to inhalers | 1 year
  Changes in therapeutic adherence of patients to inhalers with the "Inhaler Adhesion Test"

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau. Carrer Mas Casanovas 90., Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share IPD is undecided

REFERENCES:
- [Result] Partridge MR, van der Molen T, Myrseth SE, Busse WW. Attitudes and actions of asthma patients on regular maintenance therapy: the INSPIRE study. BMC Pulm Med. 2006 Jun 13;6:13. doi: 10.1186/1471-2466-6-13. PMID 16772035
- [Result] Olaguibel JM, Quirce S, Julia B, Fernandez C, Fortuna AM, Molina J, Plaza V; MAGIC Study Group. Measurement of asthma control according to Global Initiative for Asthma guidelines: a comparison with the Asthma Control Questionnaire. Respir Res. 2012 Jun 22;13(1):50. doi: 10.1186/1465-9921-13-50. PMID 22726416
- [Result] Price D, Fletcher M, van der Molen T. Asthma control and management in 8,000 European patients: the REcognise Asthma and LInk to Symptoms and Experience (REALISE) survey. NPJ Prim Care Respir Med. 2014 Jun 12;24:14009. doi: 10.1038/npjpcrm.2014.9. PMID 24921985
- [Result] Di Marco F, Verga M, Santus P, Giovannelli F, Busatto P, Neri M, Girbino G, Bonini S, Centanni S. Close correlation between anxiety, depression, and asthma control. Respir Med. 2010 Jan;104(1):22-8. doi: 10.1016/j.rmed.2009.08.005. Epub 2009 Sep 4. PMID 19733042
- [Result] Heaney LG, Conway E, Kelly C, Gamble J. Prevalence of psychiatric morbidity in a difficult asthma population: relationship to asthma outcome. Respir Med. 2005 Sep;99(9):1152-9. doi: 10.1016/j.rmed.2005.02.013. Epub 2005 Mar 23. PMID 16085217
- [Result] Ji Z, Lopez-de-Andres A, Jimenez-Garcia R, Maestre-Miquel C, Zamorano-Leon JJ, Scarano-Pereira JP, Fuentes-Alonso M, Giron-Matute WI, de Miguel-Diez J. Mental health in patients with asthma: A population-based case-control study. Respir Med. 2022 Mar;193:106758. doi: 10.1016/j.rmed.2022.106758. Epub 2022 Jan 31. PMID 35123357
- [Result] Wisnivesky JP, Lorenzo J, Feldman JM, Leventhal H, Halm EA. The relationship between perceived stress and morbidity among adult inner-city asthmatics. J Asthma. 2010 Feb;47(1):100-4. doi: 10.3109/02770900903426989. PMID 20100028
- [Result] Janssens T, Verleden G, De Peuter S, Van Diest I, Van den Bergh O. Inaccurate perception of asthma symptoms: a cognitive-affective framework and implications for asthma treatment. Clin Psychol Rev. 2009 Jun;29(4):317-27. doi: 10.1016/j.cpr.2009.02.006. Epub 2009 Mar 4. PMID 19285771
- [Result] Martinez-Moragon E, Perpina M, Belloch A, de Diego A. [Prevalence of hyperventilation syndrome in patients treated for asthma in a pulmonology clinic]. Arch Bronconeumol. 2005 May;41(5):267-71. doi: 10.1016/s1579-2129(06)60221-8. Spanish. PMID 15919008
- [Result] Veidal S, Jeppegaard M, Sverrild A, Backer V, Porsbjerg C. The impact of dysfunctional breathing on the assessment of asthma control. Respir Med. 2017 Feb;123:42-47. doi: 10.1016/j.rmed.2016.12.008. Epub 2016 Dec 18. PMID 28137495
- [Result] Sedeh FB, Von Bulow A, Backer V, Bodtger U, Petersen US, Vest S, Hull JH, Porsbjerg C. The impact of dysfunctional breathing on the level of asthma control in difficult asthma. Respir Med. 2020 Mar;163:105894. doi: 10.1016/j.rmed.2020.105894. Epub 2020 Feb 8. PMID 32056838
- [Result] Bruton A, Lee A, Yardley L, Raftery J, Arden-Close E, Kirby S, Zhu S, Thiruvothiyur M, Webley F, Taylor L, Gibson D, Yao G, Stafford-Watson M, Versnel J, Moore M, George S, Little P, Djukanovic R, Price D, Pavord ID, Holgate ST, Thomas M. Physiotherapy breathing retraining for asthma: a randomised controlled trial. Lancet Respir Med. 2018 Jan;6(1):19-28. doi: 10.1016/S2213-2600(17)30474-5. Epub 2017 Dec 14. PMID 29248433
- [Result] O'Connor E, Patnode CD, Burda BU, Buckley DI, Whitlock EP. Breathing Exercises and/or Retraining Techniques in the Treatment of Asthma: Comparative Effectiveness [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2012 Sep. Report No.: 12-EHC092-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK109355/ PMID 23101047
- [Result] Freitas DA, Holloway EA, Bruno SS, Chaves GS, Fregonezi GA, Mendonca KP. Breathing exercises for adults with asthma. Cochrane Database Syst Rev. 2013 Oct 1;(10):CD001277. doi: 10.1002/14651858.CD001277.pub3. PMID 24085551
- [Result] Prem V, Sahoo RC, Adhikari P. Comparison of the effects of Buteyko and pranayama breathing techniques on quality of life in patients with asthma - a randomized controlled trial. Clin Rehabil. 2013 Feb;27(2):133-41. doi: 10.1177/0269215512450521. Epub 2012 Jul 26. PMID 22837543
- [Result] Usmani ZA, Carson KV, Heslop K, Esterman AJ, De Soyza A, Smith BJ. Psychological therapies for the treatment of anxiety disorders in chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2017 Mar 21;3(3):CD010673. doi: 10.1002/14651858.CD010673.pub2. PMID 28322440
- [Result] Pbert L, Madison JM, Druker S, Olendzki N, Magner R, Reed G, Allison J, Carmody J. Effect of mindfulness training on asthma quality of life and lung function: a randomised controlled trial. Thorax. 2012 Sep;67(9):769-76. doi: 10.1136/thoraxjnl-2011-200253. Epub 2012 Apr 27. PMID 22544892
- [Result] Kraemer KM, McLeish A. Evaluating the role of mindfulness in terms of asthma-related outcomes and depression and anxiety symptoms among individuals with asthma. Psychol Health Med. 2019 Feb;24(2):155-166. doi: 10.1080/13548506.2018.1529326. Epub 2018 Oct 4. PMID 30286606
- [Result] Shi L, Liang D, Gao Y, Huang J, Nolan C, Mulvaney A, Poole T, Zhang H. Mindfulness and asthma symptoms: A study among college students. J Asthma. 2018 Jan;55(1):101-105. doi: 10.1080/02770903.2017.1306545. Epub 2017 May 1. PMID 28459349
- [Result] Lopez-Lois B, Gonzalez-Barcala FJ, Facal D. Application of mindfulness techniques in patients with asthma or COPD. J Asthma. 2021 Sep;58(9):1237-1246. doi: 10.1080/02770903.2020.1776729. Epub 2020 Jun 12. PMID 32475186
- [Result] Huberty J, Green J, Glissmann C, Larkey L, Puzia M, Lee C. Efficacy of the Mindfulness Meditation Mobile App "Calm" to Reduce Stress Among College Students: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jun 25;7(6):e14273. doi: 10.2196/14273. PMID 31237569
- [Result] Fazia T, Bubbico F, Nova A, Riggi E, Caimi G, Calgan B, Salvato G, Bruno S, Bottini G, Bernardinelli L. Online Short-Term Mindfulness-Based Intervention During COVID-19 Quarantine in Italy: Effects on Wellbeing, Stress, and Anxiety. Front Psychol. 2022 Jul 4;13:914183. doi: 10.3389/fpsyg.2022.914183. eCollection 2022. PMID 35859847
- [Result] Devillers-Reolon L, Mascret N, Sleimen-Malkoun R. Online Mindfulness Intervention, Mental Health and Attentional Abilities: A Randomized Controlled Trial in University Students During COVID-19 Lockdown. Front Psychol. 2022 Jul 7;13:889807. doi: 10.3389/fpsyg.2022.889807. eCollection 2022. PMID 35874414
- [Result] Vega JM, Badia X, Badiola C, Lopez-Vina A, Olaguibel JM, Picado C, Sastre J, Dal-Re R; Covalair Investigator Group. Validation of the Spanish version of the Asthma Control Test (ACT). J Asthma. 2007 Dec;44(10):867-72. doi: 10.1080/02770900701752615. PMID 18097865
- [Result] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Result] van Dixhoorn J, Duivenvoorden HJ. Efficacy of Nijmegen Questionnaire in recognition of the hyperventilation syndrome. J Psychosom Res. 1985;29(2):199-206. doi: 10.1016/0022-3999(85)90042-x. PMID 4009520
- [Result] Cooper S, Oborne J, Newton S, Harrison V, Thompson Coon J, Lewis S, Tattersfield A. Effect of two breathing exercises (Buteyko and pranayama) in asthma: a randomised controlled trial. Thorax. 2003 Aug;58(8):674-9. doi: 10.1136/thorax.58.8.674. PMID 12885982
- [Result] Slader CA, Reddel HK, Spencer LM, Belousova EG, Armour CL, Bosnic-Anticevich SZ, Thien FC, Jenkins CR. Double blind randomised controlled trial of two different breathing techniques in the management of asthma. Thorax. 2006 Aug;61(8):651-6. doi: 10.1136/thx.2005.054767. Epub 2006 Mar 3. PMID 16517572
- [Result] Fortuna AM, Feixas T, Casan P. [Measurement of fraction of exhaled nitric oxide with the portable NIOX-MINO monitor in healthy adults]. Arch Bronconeumol. 2007 Mar;43(3):176-9. doi: 10.1016/s1579-2129(07)60044-5. Spanish. PMID 17386196
- [Result] Report on skin test standardization. The Committee on Skin Test Standardization of The Netherlands Society of Allergology. Clin Allergy. 1988 May;18(3):305-10. PMID 3396198
- [Result] Juniper EF, Guyatt GH, Cox FM, Ferrie PJ, King DR. Development and validation of the Mini Asthma Quality of Life Questionnaire. Eur Respir J. 1999 Jul;14(1):32-8. doi: 10.1034/j.1399-3003.1999.14a08.x. PMID 10489826
- [Result] Sanjuas C, Alonso J, Sanchis J, Casan P, Broquetas JM, Ferrie PJ, Juniper EF, Anto JM. [The quality-of-life questionnaire with asthma patients: the Spanish version of the Asthma Quality of Life Questionnaire]. Arch Bronconeumol. 1995 May;31(5):219-26. doi: 10.1016/s0300-2896(15)30927-3. Spanish. PMID 7788083
- [Result] Plaza V, Fernandez-Rodriguez C, Melero C, Cosio BG, Entrenas LM, de Llano LP, Gutierrez-Pereyra F, Tarragona E, Palomino R, Lopez-Vina A; TAI Study Group. Validation of the 'Test of the Adherence to Inhalers' (TAI) for Asthma and COPD Patients. J Aerosol Med Pulm Drug Deliv. 2016 Apr;29(2):142-52. doi: 10.1089/jamp.2015.1212. Epub 2015 Jul 31. PMID 26230150